CLINICAL TRIAL: NCT03967067
Title: Risk Factors for Major Complications After Liver Resection: Audit of a Non-Eastern/Non-Western Experience
Brief Title: Risk Factors for Major Complications After Liver Resection
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: LiverResection
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Liver Diseases
Keywords: Audit; Liver resection; Surgical complications; non-Eastern/non-Western; Quality improvement
MeSH Terms: conditions — Liver Diseases | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: liver resection — Open or laparoscopic, major or minor hepatectomy performed using the clamp-crush technique and intermittent clamping of hepatic pedicle

SUMMARY:
The aim of this study is to determine the risk factors for major complications following liver resection in the setting of a general surgery-teaching department in Morocco, North Africa

DETAILED DESCRIPTION:
Over the past 20 years, the refinement of liver surgery techniques, anesthesiology and perioperative management has dramatically improved the safety of liver resection patients. It has also led to a concomitant extension of indications for a growing number of patients with complex benign or malignant hepatobiliary diseases and/or high risk surgeries.

Published complication rates and risk prediction models and recommendations for patients undergoing liver resection primarily stem from far East or Western high-volume specialized centers. In developing countries, including those in North Africa, specific constraints (e.g., endemic indications, such as liver cystic hydatidosis, blood shortage, and the scarcity of liver surgeons and intensive care providers) may impact liver resection outcomes but they are rarely addressed in the literature.

The aim of this study was to determine the risk factors for major complications following liver resection in the setting of a general surgery-teaching department in Morocco, North Africa

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent an hepatectomy
* between january 2010 and December 2015

Exclusion Criteria:

* All patient who only underwent liver biopsy with no resection
* Patients non operated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient who underwent a liver resection in a sugical hepatobiliary department and who had underwent preoperative serum tests, imaging workup and multidisciplinary discussion, according to the indication for LR. Adequate imaging assessment included the calculation of the future remnant liver volume (RLV) using free software, as needed. Preoperative portal embolization or a 2-step approach, including ALPPS, was considered in non-cirrhotic cases with a RLV to body weight ratio <0.5%
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
90-day Mortality rate | 90 days from surgery
  Death within 90 days of surgical procedure
90-day Complication rate | 90 days from surgery
  Defined by Clavien-Dindo grade I to IV within90 days of surgical procedure

SECONDARY OUTCOMES:
Risk factor of major complication at 90-day | 90 days from surgery
  defined by multivariate logistic regression of 90 day complication with Clavien-Dindo more than grade III

CONTACTS AND LOCATIONS:
Overall Officials: Abdelkader Belkouchi, MD, Study Director — Surgical department A Ibn Sina
Locations (1):
- Ibn Sina Hospital, Surgical department A, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dokmak S, Fteriche FS, Borscheid R, Cauchy F, Farges O, Belghiti J. 2012 Liver resections in the 21st century: we are far from zero mortality. HPB (Oxford). 2013 Nov;15(11):908-15. doi: 10.1111/hpb.12069. Epub 2013 Mar 6. PMID 23461811
- [Background] Lim C, Dejong CH, Farges O; e-HPBchir Study Group from the Association de Chirurgie Hepato-Biliaire et de Transplantation (ACHBT) (Association of Hepatobilary and Transplant Surgery). Improving the quality of liver resection: a systematic review and critical analysis of the available prognostic models. HPB (Oxford). 2015 Mar;17(3):209-21. doi: 10.1111/hpb.12346. Epub 2014 Oct 17. PMID 25322917
- [Background] Benkabbou A, Souadka A, Serji B, Hachim H, Mohsine R, Ifrine L, Belkouchi A, El Malki HO. Changing paradigms in the surgical management of cystic liver hydatidosis improve the postoperative outcomes. Surgery. 2016 Apr;159(4):1170-80. doi: 10.1016/j.surg.2015.10.029. Epub 2015 Dec 31. PMID 26747223
- [Background] Galun DA, Bulajic P, Zuvela M, Basaric D, Ille T, Milicevic MN. Is there any benefit from expanding the criteria for the resection of hepatocellular carcinoma in cirrhotic liver? Experience from a developing country. World J Surg. 2012 Jul;36(7):1657-65. doi: 10.1007/s00268-012-1544-x. PMID 22395347
- [Background] Mann CD, Palser T, Briggs CD, Cameron I, Rees M, Buckles J, Berry DP. A review of factors predicting perioperative death and early outcome in hepatopancreaticobiliary cancer surgery. HPB (Oxford). 2010 Aug;12(6):380-8. doi: 10.1111/j.1477-2574.2010.00179.x. PMID 20662788